CLINICAL TRIAL: NCT06003205
Title: Assessment of Contributing Factors to Local Bioimpedance Spectroscopy Using a Wearable Sensor: An Intervention Study
Brief Title: Contributing Factors to Local Bioimpedance Spectroscopy
Acronym: COBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mode Sensors AS (Industry)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DOC1040A COBI
Record Dates: First submitted 2023-08-02; First posted 2023-08-21 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Fluid and Electrolyte Imbalance; Overhydration; Edema
Keywords: Hydration
MeSH Terms: conditions — Water Intoxication; Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wearable bioimpedance sensor (Other): All subjects will use the investigational device and undergo several interventions: lower body negative pressure (3-40 minutes at 30 mmHg), posture intervention, and pressure intervention.
  Interventions: Device: Wearable bioimpedance sensor

INTERVENTIONS:
Device: Wearable bioimpedance sensor — The investigational device is an electronic bioimpedance-based, body-worn, battery-powered sensor intended to monitor changes in fluid volume. It is designed as an adhesive patch with four integrated electrodes.

SUMMARY:
This is an exploratory interventional study. The aim of the investigation is to identify and quantify contributing factors to local bioimpedance spectroscopy (BIS) measured by a wearable sensor patch, particularly the effect of fluid shifts caused by postural changes and lower body negative pressure (LBNP).

DETAILED DESCRIPTION:
The investigational devices (patches) will perform near-continuous measurements of multifrequency bioimpedance (BIS), temperature, and body orientation (accelerometer) during the entire period of wear (2 days). Patches will be mounted at the upper body (back and thorax) and calf. The primary objective is to assess the effect of prolonged lower body negative pressure (LBNP) on the BIS of the calf. The target population is healthy volunteers between 18-50 years old.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 50 years of age, at the time of signing the informed consent
* Overtly healthy as determined by medical evaluation including medical history, physical examination and focused cardiac ultrasound.
* Use of adequate birth control for women of childbearing potential. Inclusion is possible when an acceptable effective contraceptive measure is used (combined (estrogen and progestogen containing) hormonal contraception, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner or sexual abstinence).
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Known allergies or skin sensitivities to electrode hydrogel and/or acrylic adhesives
* Breached skin at patch mounting area.
* Implantable pulse generators such as pacemakers and defibrillators, and/or use of other electrical medical equipment for which an interaction effect with the investigational device cannot be ruled out.
* Planned magnetic resonance (MR) imaging during the investigation period
* Any medical condition limiting physical exertional capacity or requiring regular medication (allergy and contraceptives excepted).
* Pregnancy
* Breastfeeding
* History of syncope (syncope of presumed vasovagal nature with known precipitating factor excepted).
* Any known cardiac disease that, at the investigator's discretion, warrants exclusion from the study, including but not limited to cardiac arrhythmia, esophageal varices, and aneurysms.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Relative change in extracellular resistance of the calf from t0 to t1 (immediately before and after 40 minutes of LBNP at 30 mmHg), measured by the investigational bioimpedance device | 40 minutes
  Relative change in extracellular resistance at the calf from before to after 40 minutes of lower body negative pressure, to assess the effect of prolonged LBNP.

SECONDARY OUTCOMES:
Change in extracellular resistance at the upper back following postural changes, measured by the investigational bioimpedance device. | 6 hours
  Relative change in extracellular resistance at the upper back following changes in posture
Changes in extracellular resistance at the upper back following application of three different external pressures. | 2 hours
  Mean differences in extracellular resistance of the upper back, when the subject lays in a supine position on three different surfaces. Extracellular resistance is measured by the investigational bioimpedance device.
Frequency and severity of adverse device effects | 3 days
  To assess the safety of the investigational device in healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Sigve N Aas, PhD, Study Director — Mode Sensors AS; Lars Ø Høiseth, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Physiology lab. Aker hospital, Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No